CLINICAL TRIAL: NCT00523276
Title: Immune Responses, Transmission and Nucleotide Polymorphisms in Families With SARS Virus Infections
Brief Title: SARS Survivor Evaluations
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 06-0048
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Coronavirus (SARS-CoV)
Keywords: Severe acute respiratory syndrome, SARS, China
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Sera, PBMCs

GROUPS / COHORTS (3):
- HCWs: Who may/may not have contact with SARS patients
- Family/close contacts: No illness but household/close contact
- SARS subjects: Diagnosed with active disease

SUMMARY:
The purpose of this study is to understand how severe acute respiratory syndrome (SARS) spreads within families, if significant disease resulted, and how the body responds to SARS. The study will also explore the affects of SARS on genetics and the immune system (the body system that fights disease). Up to 1000 people residing in Beijing, China may be involved in this study. Adult survivors of SARS (numbering 200) and their family members including children age 4 and up will be asked to participate in the study. The study will recruit an additional 200 persons, who will be matched with SARs survivors of similar age, gender, health status, and housing/work location, and recruited as comparators. Blood will be taken from all volunteers and tested for the presence of SARS antibodies (proteins made by the body's immune system in response to something that can cause infection). Health and clinic/hospital visit records may be reviewed.

DETAILED DESCRIPTION:
This study will investigate immune responses, transmission and nucleotide polymorphisms in families with severe acute respiratory syndrome (SARS) virus infections. Study objectives are to: develop an immune response profile to SARS coronavirus (SARS CoV) among SARS survivors; ascertain whether there was spread of SARS CoV within the family and whether significant disease resulted; and determine whether 1 or more nucleotide polymorphisms relate to occurrence and severity of SARS CoV disease or immunologic responses. Up to 1,000 persons residing in Beijing, China, will participate in this study and will include the following groups: 200 adult (greater than or equal to18 years of age) subjects, previously experiencing SARS caused by SARS Coronavirus; their household/family members, including children ages 4 and up (male or female); and an additional 200 adults matched for characteristics (age, gender, health status and housing/work location) of the 200 SARS survivors. As much as possible (for DNA tests), these controls will be persons involved in health care with a possible SARS exposure during the epidemic. Blood will be obtained from all subjects and used for SARS CoV antibody assays. Additional studies will be performed with blood specimens from selected subjects. Tests for serum antibodies will be used to identify infected persons in each family. For any who possess specific antibodies, a review of their health and clinic/hospital visit records for the SARS epidemic period will be conducted to identify any illness, its type and severity. A control for interpretation can be illnesses during the study period in uninfected family members. Data will be analyzed by age, gender, and health status of family members, the severity of SARS illness in the index case and the time of return to the home environment. The illness data will be obtained from medical records and not from subject memory. To assess health status, subjects for this study will have a chest x-ray performed and 15 mL of blood obtained for complete blood counts, liver function, to include ALT, and creatinine. For study purposes, 30 to 100 mL of blood will be collected from SARS survivors and from 50 matched controls (age, gender and health status). Illnesses from medical records will be characterized for severity and will include extent of x-ray changes, need for oxygen therapy, medical care in the intensive care unit and extent of leukocyte changes. Microarray chips that contain human genes determining immune responses, production of cytokines and chemokines and a number of other potential responses to illness have been constructed. PureGene kits will be provided for isolation of DNA from blood specimens for testing for polymorphisms. These analyses will be performed on the 200 SARS survivors, the 200 matched controls and on family members. The DNA samples will be shipped to laboratories at Baylor College of Medicine for analysis using the microarray chips.

ELIGIBILITY:
Inclusion Criteria:

Severe Acute Respiratory Syndrome (SARS) Survivors and Controls:

1. An adult (>= 18 years of age) proven in hospital/laboratory records to have had SARS as defined by the World Health Organization
2. A control matched for age, gender and health status similar to a SARS survivor and with a possible SARS exposure (healthcare personnel).
3. Granting informed consent

Family Members of SARS Survivors:

1. Family members currently age 4 or older who were living in a household with the SARS survivor study case at the time of SARS occurrence.
2. Informed consent granted by subject or parent if child is less than 18 years old.

Exclusion Criteria:

Severe Acute Respiratory Syndrome (SARS) Survivors and Controls:

1. Presence of an acute illness.
2. Hemoglobin below normal range for gender and age.
3. Current pregnancy or possible pregnancy (by history).

Family Members of SARS Survivors:

1. Current pregnancy or possible pregnancy (by history).

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult (> 18 yo) SARS survivors and family members. Adult matched controls
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Positive serology, SARS CoV | at time of assay

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Beijing You'An Hospital, Beijing, Beijing Municipality